CLINICAL TRIAL: NCT00190125
Title: The Influences of Malnutrition and Inflammation Complex Syndrome in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: National Taiwan University (Other)
Other Study IDs: FEMH-94008
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2005-08

CONDITIONS: Hemodialysis; Malnutrition; Inflammation; Myocardial Ischemia; Cerebrovascular Accident
Keywords: Hemodialysis; Malnutrition; Inflammation
MeSH Terms: conditions — Malnutrition; Inflammation; Myocardial Ischemia; Stroke

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to explore the severity of malnutrition and inflammation in Taiwanese hemodialysis patients.

DETAILED DESCRIPTION:
Cardiovascular disease is the major of cause of mortality of hemodialysis patients. In addition to diabetes and hypertension, malnutrition and chronic inflammation are well-known to be major risk factors of cardiovascular diseases in normal population. For detecting the malnutrition and chronic inflammation and understanding the exact influences to hemodialysis patients, we conduct this study. We will collect the biochemical parameters, inflammatory markers, lipid parameters, hematologic parameters, and genomic DNA of patients. Then we will prospectively record the hospitalization, cardiovascular events, complications of arteriovenous fistula/graft, and mortality. According to the above results, we try to explore the exact role of malnutrition and inflammation in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received hemodialysis therapy for more than three months

Exclusion Criteria:

* Having active infection diseases now
* Patients who have a malignancy
* Had cardiovascular events in recent three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Study Completion 2007-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Sen Peng, M.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Pan-Chiao, Taipei Country, Taiwan

REFERENCES:
- [Background] Kalantar-Zadeh K, Ikizler TA, Block G, Avram MM, Kopple JD. Malnutrition-inflammation complex syndrome in dialysis patients: causes and consequences. Am J Kidney Dis. 2003 Nov;42(5):864-81. doi: 10.1016/j.ajkd.2003.07.016. PMID 14582032
- [Background] Kalantar-Zadeh K, Kopple JD, Block G, Humphreys MH. Association among SF36 quality of life measures and nutrition, hospitalization, and mortality in hemodialysis. J Am Soc Nephrol. 2001 Dec;12(12):2797-2806. doi: 10.1681/ASN.V12122797. PMID 11729250
- [Background] Kalantar-Zadeh K, McAllister CJ, Lehn RS, Lee GH, Nissenson AR, Kopple JD. Effect of malnutrition-inflammation complex syndrome on EPO hyporesponsiveness in maintenance hemodialysis patients. Am J Kidney Dis. 2003 Oct;42(4):761-73. doi: 10.1016/s0272-6386(03)00915-6. PMID 14520627
- [Background] Kalantar-Zadeh K, Block G, McAllister CJ, Humphreys MH, Kopple JD. Appetite and inflammation, nutrition, anemia, and clinical outcome in hemodialysis patients. Am J Clin Nutr. 2004 Aug;80(2):299-307. doi: 10.1093/ajcn/80.2.299. PMID 15277149
- [Background] Kalantar-Zadeh K, Mehrotra R, Fouque D, Kopple JD. Metabolic acidosis and malnutrition-inflammation complex syndrome in chronic renal failure. Semin Dial. 2004 Nov-Dec;17(6):455-65. doi: 10.1111/j.0894-0959.2004.17606.x. PMID 15660576